CLINICAL TRIAL: NCT02734823
Title: Long Term Effects of Tyrosine Kinase Inhibitors on Ovarian Reserve and Fertility, A Pilot Study
Brief Title: Long Term Effects of Tyrosine Kinase Inhibitor Therapy on Ovarian Reserve and Fertility in Patients With Chronic Myeloid Leukemia or Gastrointestinal Stromal Tumor
Status: Withdrawn | Type: Observational
Why Stopped: Lack of accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-15-7; NCI-2016-00352 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-15-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Gastrointestinal Stromal Tumor; Premenopausal
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (ovary imaging, hormonal analysis): Patients undergo transvaginal ultrasound for antral follicles analysis and collection of serum for ovarian reserve markers and hormonal analysis before TKI therapy and at 12, 24, and 48 weeks.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Procedure: Ultrasonography

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of serum
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Procedure: Ultrasonography — Undergo transvaginal pelvic ultrasonography
  Other Names: ULTRASOUND; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This pilot research trial studies the long term effects of tyrosine kinase inhibitor therapy on ovarian reserve and fertility in patients with chronic myeloid leukemia or gastrointestinal stromal tumor. Studying ovary imaging, ovarian reserve markers, and hormone levels from patients receiving tyrosine kinase inhibitor therapy may help doctors learn more about the effects of tyrosine kinase inhibitor therapy on ovarian function and fertility.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect preliminary information to help design a study to look at longitudinal changes in markers of ovarian reserve and menstruation in premenopausal women undergoing tyrosine kinase inhibitors (TKI) therapy.

SECONDARY OBJECTIVES:

I. Evaluate ovarian response to controlled ovarian hyperstimulation in patients who elect to undergo in vitro fertilization (IVF) for fertility preservation.

OUTLINE:

Patients undergo transvaginal ultrasound for antral follicles analysis and collection of serum for ovarian reserve markers and hormonal analysis before TKI therapy and at 12, 24, and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic myeloid leukemia (CML), gastrointestinal stromal tumor (GIST), non metastatic cancer where TKI is the first line agent
* Premenopausal (has had menses at any time in the preceding 12 consecutive months)
* Has not undergone a hysterectomy or bilateral oophorectomy
* Willing to use non-hormonal (ie: barrier method or abstinence) as form of contraception during the one year of study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy in the past
* Patients may not be receiving any other investigational agents
* Patients must not be pregnant or nursing
* Other medical conditions or treatments that affect hormonal levels (potentially confounding interpretation of results)
* Patients with ongoing hormonal contraception or unwilling or unable to discontinue will not eligible

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with chronic myeloid leukemia or gastrointestinal stromal tumor undergoing TKI therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2024-03-14 (Estimated); Study Completion 2024-03-14 (Estimated)

PRIMARY OUTCOMES:
Changes in markers of ovarian reserve in premenopausal women undergoing tyrosine kinase inhibitor therapy for cancer | Baseline to up to 1 year
  Standard descriptive statistics and scatter plots will be used to summarize patterns by cohorts at each time point. Regression methods will be used to render data compatible with the assumption of the normal distribution. Analysis will be undertaken to obtain preliminary estimates of ovarian reserve over time and to elucidate whether TKI therapy produces a clinically meaningful change in ovarian reserve marker.

SECONDARY OUTCOMES:
Ovarian response to controlled ovarian hyperstimulation in patients who elect to undergo IVF for fertility preservation | Up to 1 year
  The results of their stimulation protocol will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Woo, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States